CLINICAL TRIAL: NCT01969513
Title: Effectiveness of the Epley Manoeuvre Performed in Primary Care to Treat Posterior Canal Benign Paroxysmal Positional Vertigo
Brief Title: Effectiveness of the Epley Manoeuvre Performed in Primary Care to Treat Benign Paroxysmal Positional Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other); Red Española de Atención Primaria (REAP) (Unknown); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4R13/029-1; ID: 4R13/017
Record Dates: First submitted 2013-03-27; First posted 2013-10-25 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Benign Positional Paroxysmal Vertigo
Keywords: Vestibular Diseases; Vertigo; Primary care; Epley maneuver
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vestibular Diseases; Vertigo

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INTERVENTION ARM (Experimental): Patients meeting the inclusion criteria will be randomly assigned to the experimental group. They will receive Epley's manoeuvre plus betahistine 8mg three times a day until they no longer have symptoms. The Epley's manoeuvre will be performed only on the first visit.
  Interventions: Procedure: PROCEDURE: EPLEY MANOEUVRE
- CONTROL GROUP (Sham Comparator): Patients meeting the inclusion criteria will be randomly assigned to the control group. These patients will receive sham manoeuvre (simulated Epley manoeuvre) plus betahistine 8mg three times a day until they no longer have symptoms. Placebo manoeuvre is performed with the patient lying down over the affected side for 5 minutes as it is described in similar studies.
  Interventions: Procedure: PROCEDURE: SHAM MANOEUVRE

INTERVENTIONS:
Procedure: PROCEDURE: EPLEY MANOEUVRE — The procedure involves a series of four movements of the head and body from sitting to lying, rolling over and back to sitting.
  Other Names: Canalith repositioning manoeuvre
  Arms: INTERVENTION ARM
Procedure: PROCEDURE: SHAM MANOEUVRE — Placebo manoeuvre is performed with the patient lying down over the affected side for 5 minutes as it is described in similar studies.
  Other Names: Simulated Epley manoeuvre
  Arms: CONTROL GROUP

SUMMARY:
Vertigo is a common medical issue with a broad expectrum of diagnoses that requires a global approach to patients through structured clinical interview and physical examination. The main cause of vertigo in primary care is benign paroxysmal positional vertigo (BPPV) that is confirmed by a positive Dix-Hallpike positional test and treated with repositioning manoeuvres. Objective: To evaluate the effectiveness of Epley's manoeuvre performed by general practitioners (GPs) in the treatment of BPPV. Design: randomized clinical trial conducted in primary care. Scope: Two urban centres serving about 50,000 patients. Patients: All patients with newly diagnosed BPPV will be offered to participate in the study and will be randomly assigned to the treatment group (Epley manoeuvre) or control group (sham manoeuvre) and both groups will receive betahistine. Outcome variables will be: response to the Dix Hallpike test, patients will inform if vertigo was present during the last week (dichotomous variable: yes/no), intensity of vertigo symptoms on a Likert scale in the past week, score of Vertigo Handicap Inventory and quantity of betahistine taken. Statistical analysis: Descriptive statistics of all variables collected. Groups will be compared using the intent-to-treat approach and either parametric or nonparametric tests depending on the nature and distribution of the variables. Chi-square test or exact Fisher test will be used to compare qualitative measures and Student's t test o Mann Whitney U test will be used for between-group comparison of variables.

Positive results from our study will highlight that treatment of BPPV can be performed by trained GPs and its widespread practice can greatly improve the quality of life of these patients.

DETAILED DESCRIPTION:
DESIGN:

Randomized clinical trial conducted by general practitioners (GP) who received a two hour training to perform the manoeuvres under the supervision of an otorhinolaryngologist. Patients will be reevaluated 1 week, 1 month and 1 year after the first visit by a different GP from the first visit to accomplish blinding of study participants and personnel.

MAIN OBJECTIVE:

The aim of this study is to determine whether the improvement is greater in intervention group than in control group in terms of Dix-Hallpike manoeuvre turning negative, subjective perception of vertigo and quality of life, and less amount of betahistine taken.

The main objective is the response of treatment in the second visit (1 week after the first visit), although new assessments will be carried out at day 30 and one year after the first visit.

ELIGIBILITY:
INCLUSION CRITERIA

* Patients aged 18 years and older who attend our primary care centre, with suspected diagnosis of BPPV, and present vertigo or nystagmus with DH manoeuvre. All other causes of vertigo will be ruled out.
* Written informed consent will be obtained from all subjects of both intervention group and control group prior to its inclusion in the study.

EXCLUSION CRITERIA

* Previous or current diagnoses of labyrinth's diseases such as Meniere's disease, labyrinthitis or vestibular neuronitis.
* Contraindications to canalith repositioning procedures: cervical spinal stenosis, severe kyphoscoliosis, limited cervical mobility, Down syndrome, advanced rheumatoid arthritis, cervical radiculopathies, Paget's disease, morbid obesity, ankylosing spondylitis, severe lumbar dysfunction and spinal cord injuries.
* Pregnancy or breastfeeding.
* Contraindications of betahistine.
* Refusal of patients to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
PERSISTENCE OF VERTIGO | One week after recruitment
  Evaluate if the Dix Hallpike manoeuvre produces dizziness or nystagmus to the right or left or both sides. If they are present at both sides the manoeuvre will be considered positive for the side where the symptoms are intense.

SECONDARY OUTCOMES:
BETAHISTINE TABLET COUNT | One week after recruitment
  All patients will be prescribed betahistine 8mg three times a day until they no longer have symptoms. We will analyze whether patients' self-report of the sum of betahistine tablets taken are lower in intervention group in comparison to control group
NEW EPISODES OF BENIGN PAROXYSMAL POSITIONAL VERTIGO IN THE ANNUAL VISIT | One year after recruitment
  Analyze if new episodes have occurred before the annual visit and calculate the elapsed time between the first visit and the new episode.
SEVERITY OF VERTIGO MEASURED ON A LIKERT SCALE | One year after recruitment
  Patients will be asked to rate the severity of the vertigo on a 10 point Likert scale: 0 = not experiencing, 10 = worst and unbearable.
DIZZINESS HANDICAP INVENTORY SHORT FORM (DHI-S) | One week after recruitment
  The questionnaire used is an adapted version of the original DHI into Spanish by López- Escamez. It was translated and back translated by two interpreters with clinical experience and both translations were discussed in a consensus meeting with one of the researchers yielding to an adapted version. The internal consistency coefficient, Cronbach alpha, was 0.8014.
  This 10 item self-assessment inventory will evaluate the self-perceived handicapping effects imposed by dizziness.
PATIENTS REPORTING PERSISTENCE OF VERTIGO | One week after recruitment
  Patients will inform if vertigo was present during the last week (Dichotomous variable: yes/no).
PATIENTS REPORTING PERSISTENCE OF VERTIGO | One month after recruitment
  Patients will inform if vertigo was present during the last week (Dichotomous variable: yes/no).
PATIENTS REPORTING PERSISTENCE OF VERTIGO | One year after recruitment
  Patients will inform if vertigo was present during the last week (Dichotomous variable: yes/no).
DIZZINESS HANDICAP INVENTORY SHORT FORM (DHI-S) | One month after recruitment
  The questionnaire used is an adapted version of the original DHI into Spanish by López- Escamez. It was translated and back translated by two interpreters with clinical experience and both translations were discussed in a consensus meeting with one of the researchers yielding to an adapted version. The internal consistency coefficient, Cronbach alpha, was 0.8014.
  This 10 item self-assessment inventory will evaluate the self-perceived handicapping effects imposed by dizziness.
DIZZINESS HANDICAP INVENTORY SHORT FORM (DHI-S) | One year after recruitment
  The questionnaire used is an adapted version of the original DHI into Spanish by López- Escamez. It was translated and back translated by two interpreters with clinical experience and both translations were discussed in a consensus meeting with one of the researchers yielding to an adapted version. The internal consistency coefficient, Cronbach alpha, was 0.8014.
  This 10 item self-assessment inventory will evaluate the self-perceived handicapping effects imposed by dizziness.
SEVERITY OF VERTIGO MEASURED ON A LIKERT SCALE | One month after recruitment
  Patients will be asked to rate the severity of the vertigo on a 10 point Likert scale: 0 = not experiencing, 10 = worst and unbearable.
SEVERITY OF VERTIGO MEASURED ON A LIKERT SCALE | One week after recruitment
  Patients will be asked to rate the severity of the vertigo on a 10 point Likert scale: 0 = not experiencing, 10 = worst and unbearable.
BETAHISTINE TABLET COUNT | One month after recruitment
  All patients will be prescribed betahistine 8mg three times a day until they no longer have symptoms. We will analyze whether patients' self-report of the sum of betahistine tablets taken are lower in intervention group in comparison to control group.

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Ballvé, Principal Investigator — Institut Català de la Salut
Locations (1):
- CAP Florida, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Carrillo Munoz R, Ballve Moreno JL, Villar Balboa I, Rando Matos Y, Cunillera Puertolas O, Almeda Ortega J, Rodero Perez E, Monteverde Curto X, Rubio Ripolles C, Moreno Farres N, Matos Mendez A, Gomez Nova JC, Bardina Santos M, Villarreal Minano JJ, Pacheco Erazo DL, Hernandez Sanchez AM; Grupo de estudio del vertigo en atencion primaria Florida. Disability perceived by primary care patients with posterior canal benign paroxysmal positional vertigo. BMC Fam Pract. 2019 Nov 13;20(1):156. doi: 10.1186/s12875-019-1035-3. PMID 31722671
- [Derived] Ballve Moreno JL, Carrillo Munoz R, Villar Balboa I, Rando Matos Y, Arias Agudelo OL, Vasudeva A, Bigas Aguilera O, Almeda Ortega J, Capella Guillen A, Buitrago Olaya CJ, Monteverde Curto X, Rodero Perez E, Rubio Ripolles C, Sepulveda Palacios PC, Moreno Farres N, Hernandez Sanchez AM, Martin Cantera C, Azagra Ledesma R. Effectiveness of the Epley's maneuver performed in primary care to treat posterior canal benign paroxysmal positional vertigo: study protocol for a randomized controlled trial. Trials. 2014 May 21;15:179. doi: 10.1186/1745-6215-15-179. PMID 24886338